CLINICAL TRIAL: NCT04228809
Title: Long-term Efficacy of Transcranial Direct Current Stimulation in Chronic Migraine With Medication Overuse: a Phase III, Placebo Controlled, Randomised Clinical Trial (Edisom)
Brief Title: tDCS in Chronic Migraine With Medication Overuse (Edisom)
Acronym: Edisom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Edisom
Record Dates: First submitted 2020-01-04; First posted 2020-01-14 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Migraine Disorders; Medication Overuse Headache
MeSH Terms: conditions — Migraine Disorders; Headache Disorders, Secondary | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: sham
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- anodal tDCS (Experimental): anodal tDCS stimulation
  Interventions: Device: tDCS
- cathodal tDCS (Active Comparator): cathodal tDCS stimulation
  Interventions: Device: tDCS
- sham tDCS (Placebo Comparator): sham tDCS stimulation (stopped after 30 seconds)
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — transcranial direct current stimulation

SUMMARY:
Transcranial direct current stimulation (tDCS) was suggested to provide beneficial effects in chronic migraine (CM), a condition often associated with medication overuse (MO) for which no long-term therapy is available.

DETAILED DESCRIPTION:
We conducted a randomized controlled trial to assess long-term efficacy of tDCS. Adults diagnosed with CM and MO were assigned to receive in a 1:1:1 ratio anodal, cathodal, or sham tDCS daily for five consecutive days, along with standardized drug withdrawal protocol with intravenous administration of dexamethasone 4 mg and ademetionine 200 mg in saline solution, and oral bromazepam 1.5 mg three times daily.

Primary outcome was 50% reduction of days of headache per month at 12 months. Co-secondary outcomes were 50% reduction of days of headache per month at 6 months, reduction of analgesic intake per month, and change in disability and quality of life, catastrophizing, depression, state and trait anxiety, dependence attitude and allodynia intensity. Patients were not allowed to take any migraine prophylaxis drug for the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* chronic migraine with medication overuse according to the International Headache Society criteria. Diagnosis was confirmed on the basis of a daily headache diary that all eligible patients filled out in the last month prior to the enrollment. Patients should have failed at least two prophylaxis therapies. Written informed consent.

Exclusion Criteria:

* known diagnosis of major depression or other major psychiatric disorders identified after psychiatric consultation, cardiac pace maker, clips for previous head surgery, cochlear implant, history of epilepsy, known idiopathic intracranial hypertension, harmful alcohol consumption, pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
days of headache per month (long-term) | 12 months
  no. patients with 50% reduction of days of headache per month

SECONDARY OUTCOMES:
days of headache per month (mid-term) | 6 months
  no. patients with 50% reduction of days of headache per month
analgesic intake per month | 6 and 12 months
  percentage of reduction of analgesic intake per month compared to baseline
disability | 6 and 12 months
  Migraine Disability Assessment (MIDAS). MIDAS-score
  0-:5 low disability
  6-10: MILD disability 11-20: Moderate disability more than 2:0 Severe disability.
catastrophizing attitude | 6 and 12 months
  Pain Catastrophizing Scale (PCS) pathological more than 30 (total score) no cut off for the subscales
depression | 6 and 12 months
  Beck Depression Inventory (BDI) score more than 7
state and trait anxiety | 6 and 12 months
  Spielberger questionnaires STAIY1-Y2 ; score between 20-80
dependence attitude | 6 and 12 months
  Leed questionnaire score
  Under 10: low dependency
  10-22: medium dependency
  more than 22: high dependency
allodynia intensity | 6 and 12 months
  Allodynia Symptoms Checklist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grazzi L, Usai S, Bolognini N, Grignani E, Sansone E, Tramacere I, Maravita A, Lauria G. No efficacy of transcranial direct current stimulation on chronic migraine with medication overuse: A double blind, randomised clinical trial. Cephalalgia. 2020 Oct;40(11):1202-1211. doi: 10.1177/0333102420931050. Epub 2020 Jun 14. PMID 32536270